CLINICAL TRIAL: NCT02172651
Title: Study to Identify Transcriptional Targets of Vitamin D in Patients With Stage I-III Colon Cancer or Resectable Colon Cancer Liver Metastases Receiving Preoperative Vitamin D Supplementation.
Brief Title: Vitamin D in Patients With Stage I-III Colon Cancer or Resectable Colon Cancer Liver Metastases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pharmavite LLC (Industry)
Responsible Party: Principal Investigator, Kimmie Ng, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-091; P50CA127003-06A1 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Stage, Colon Cancer; Stage I-III Colon Cancer; Stage IV Colon Cancer With Resectable Liver Metastases
Keywords: Vitamin D; Stage I-III colon cancer; Stage IV colon cancer; Resectable liver metastases
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Vitamin D3 - Blinded Registration (Experimental): One capsule of vitamin D3 10,000 IU orally once daily for 14 days until the date of surgery. To allow for some flexibility in the scheduling of surgery, patients can be treated with preoperative vitamin D3 for up to 28 days. On the morning of surgery, prior to operating, a second blood sample will be collected for follow-up 25(OH)D, calcium, and albumin determination. Colon and liver resection will occur per institutional standards of care, and malignant and adjacent benign tissue will be collected for the laboratory endpoints described in this protocol.
  Interventions: Drug: Vitamin D3
- Placebo - Blinded Registration (Placebo Comparator): One placebo capsule orally once daily for 14 days until the date of surgery. To allow for some flexibility in the scheduling of surgery, patients can be treated with preoperative placebo for up to 28 days. On the morning of surgery, prior to operating, a second blood sample will be collected for follow-up 25(OH)D, calcium, and albumin determination. Colon and liver resection will occur per institutional standards of care, and malignant and adjacent benign tissue will be collected for the laboratory endpoints described in this protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Take five 10,000 IU capsules (total 50,000 IU) once daily for 7 days, followed by one 10,000 IU capsule once daily until surgery.
  Other Names: cholecalciferol (vitamin D3)
  Arms: Vitamin D3 - Blinded Registration
Drug: Placebo — Take five placebo capsules once daily for 7 days, followed by one placebo capsule once daily until surgery.
  Arms: Placebo - Blinded Registration

SUMMARY:
This study seeks to learn more about the vitamin D receptor and its relationship to colon cancer. The Vitamin D receptor is found in colon cancer cells. When Vitamin D binds to the receptor in the cancer cells, it may stop cancer cells from growing abnormally and may cause cancer cell death. Vitamin D has been used in other research studies and information from those other research studies suggests that Vitamin D may help in the treatment of colon cancer.

Participants will receive either high-dose vitamin D or standard-dose vitamin D. The study drug will be given 14-28 days prior to your surgery. The number of days will depend on when the surgery is scheduled.

DETAILED DESCRIPTION:
The participant will be given a study drug-dosing diary to keep track of when they take the study drug. The participant will be taking the study drug once every day, for 14 - 28 days, prior to their surgery.

* Run-In Phase: The first 6-12 participants will receive high-dose vitamin D prior to surgery. The number of participants in this phase will be based on the results of the analyzed research samples.
* Randomized Phase: Because no one knows which of the study options is best, the participant will be "randomized" into one of the study groups: high dose vitamin D or standard dose vitamin D.

  * 48 Participants will be randomized to receive high-dose vitamin D or standard-dose vitamin D. Randomization means that the participants are put into a group by chance. Neither the participant nor the research doctor will choose what group the participant will be in. The participant will have an equal chance of getting assigned to each arm (like flipping a coin). The randomized phase will enroll to two groups at the same time:

    * Group A: 24 participants with a recent diagnosis of stage I, II or III colon cancer will be randomized to receive high-dose vitamin D or standard-dose vitamin D.
    * Group B: 24 participants with resectable liver metastases from colon cancer will be randomized to receive high-dose vitamin D or standard-dose vitamin D.

Additional research procedures to be performed on study:

* Blood samples will be collected for research purposes (a little more than 2 teaspoons of blood). The samples will be collected immediately prior to the participant's surgery and used to study the vitamin D receptor and pathway, as well as its relationship to colon cancer. Some of this blood will be stored to be used for future cancer research.
* Tumor tissue will be collected for research purposes at the time of the participant surgery. This tissue will also be used to study the vitamin D receptor and pathway, as well as its relationship to colon cancer. Some of the tumor tissue collected will be sent for use in a separate, but related study. In this study, the participant's tumor will be used to grow cell lines. This means the participant's tumor cells will be multiplied in the lab. These cell lines will be used to study the binding sites in the genes of participants and learn more about vitamin D's role in preventing colon cancer.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Participants must have histologically confirmed adenocarcinoma of the colon that is localized, with no evidence of distant metastasis (stage I, II, or III), and for which surgical resection of the primary tumor is being planned;

  --OR
* Participants must have histologically or cytologically confirmed adenocarcinoma of the colon with resectable liver metastases for which liver resection is being planned.
* No prior radiation therapy or systemic treatment is allowed for patients undergoing resection of stage I, II, or III colon cancer.
* Prior systemic treatment or radiation therapy is allowed for patients with resectable liver metastases.

  * The last dose of chemotherapy or radiation must have been administered at least 4 weeks prior to liver surgery.
  * The last dose of bevacizumab must have been administered at least 6 weeks prior to liver resection.
* Age ≥18 years.
* ECOG performance status ≤ 1 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * Total bilirubin ≤1.5× institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN, or <5x ULN if clearly attributable to liver metastases
  * Serum calcium (corrected for albumin level) ≤ 1x institutional ULN
  * Serum creatinine within normal institutional limits or creatinine clearance ≥60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Participants on full-dose anticoagulation are eligible if the following criteria are met:

  * Participant has an in-range INR (usually 2-3) on a stable dose of warfarin or is on a stable dose of low molecular weight heparin
  * Participant has no active bleeding or pathological condition that carries a high risk of bleeding (i.e., tumor involving major vessels or known varices)
  * Participants receiving anti-platelet agents are eligible. In addition, patients who are on daily prophylactic aspirin or anticoagulation for atrial fibrillation are eligible.
  * Discontinuation of anticoagulation, aspirin, and/or anti-platelet agents prior to surgery will occur according to institutional standards of care.
* Non-pregnant and not nursing

  * Women of child-bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 14 days prior to study entry. Women of child-bearing potential include any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ≥12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone level >35 mIU/mL). Women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child-bearing potential.
  * The effects of higher-dose vitamin D3 and colon or liver surgery (and associated perioperative medications and anesthesia) on the developing human fetus are unknown and may pose unacceptable risk. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Prior systemic therapy, radiotherapy, or investigational agent in participants undergoing surgery for stage I, II, or III colon cancer.
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for bevacizumab) of liver resection.
* Concurrent use of other anti-cancer therapy, including chemotherapy agents, targeted agents, biological agents, immunotherapy, or investigational agents not otherwise specified in this protocol.
* Inability to swallow pills.
* History of malabsorption or uncontrolled vomiting or diarrhea, or any other disease significantly affecting gastrointestinal function that could interfere with absorption of oral medications.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vitamin D.
* Regular use of supplemental vitamin D totaling ≥ 2,000 IU/day in the past year.

  * Use of supplemental vitamin D or supplements containing vitamin D beyond the protocol-prescribed study treatment is not allowed during the treatment period of this clinical trial.
  * In order to maintain blinding, vitamin D levels should not be routinely checked at screening or during the study by the treating investigator. Vitamin D levels will be assayed only as part of the research blood samples collected during the study. If there are concerns related to a participant's vitamin D status, the lead Principal Investigator should be contacted for further discussion.
* Use of chronic oral corticosteroid therapy, lithium, phenytoin, quinidine, isoniazid, and/or rifampin (all of which can cause vitamin D depletion). Short-term use of corticosteroids as anti-emetic therapy for chemotherapy is permitted.
* Regular use of thiazide diuretics (i.e., hydrochlorothiazide), which can lead to hypercalcemia, and unwillingness or inability to discontinue or switch to an alternative anti-hypertensive agent.
* Pre-existing hypercalcemia (defined as baseline serum calcium above the institutional ULN, corrected for albumin level if albumin is not within institutional limits of normal).

  -- The use of supplemental calcium or supplements containing calcium is prohibited during the treatment period of this clinical trial.
* Known active hyperparathyroid disease or other serious disturbance of calcium metabolism in the past 5 years.
* History of symptomatic genitourinary stones within the past year.
* Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, may increase the risks associated with study participation or study treatment, limit compliance with study requirements, or interfere with the interpretation of study results.
* Pregnant or nursing women or men/women of child-bearing potential who are unwilling to employ adequate contraception.

  -- Pregnant and nursing women are excluded from this study because there is an unknown but potential risk of adverse events related to higher-dose vitamin D3 and colon or liver surgery (and associated perioperative medications and anesthesia) on the human fetus. Consequently, breastfeeding should be discontinued if the mother is enrolled on the study.
* History of prior or synchronous malignancy except:

  * A malignancy that was treated with curative intent, for which there has been no known active disease for >3 years prior to randomization, and for which the risk of recurrence is low as determined by the investigator.
  * Curatively treated non-melanoma skin malignancy, cervical cancer in situ, or prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Known positive test for human immunodeficiency virus (HIV), hepatitis C virus, or acute or chronic hepatitis B infection.

  * Participants with these infections are ineligible because they are at increased risk of significant complications in the perioperative period, particularly for active hepatitis B or C patients undergoing liver resection. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-07-14 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
VDR Binding Sites | 14 to 28 days
  For patients undergoing primary colon resection, the goal is to identify VDR binding sites in malignant and normal colonic tissue collected from colon cancer patients treated with high-dose vitamin D3 versus placebo.
  ChIP-Seq will be performed on frozen tumor tissue and adjacent normal colon tissue to determine VDR binding sites, which will be compared between the high-dose vitamin D and placebo arms, and between malignant tumor and normal colon tissue.

SECONDARY OUTCOMES:
Changes in TME | 14 to 28 days
  For patients undergoing liver resection, the goal is to characterize changes in the TME of liver metastases collected from colon cancer patients treated with high-dose vitamin D3 versus placebo.
  Tumor microarrays will be constructed from FFPE tissue to evaluate the densities and co-localization of TILs and other immune cell types with tumor epithelial cells using custom multiplex immunofluorescence assays with supervised machine learning. A custom vitamin D-immune panel will also be used to measure nuclear VDR and cytoplasmic CYP27B1 expression at the single cell level in pan-CK+ tumor epithelial cells, numerous immune cell populations (CD3+CD4+ T helper cells, CD3+CD8+ cytotoxic T cells, CD68/CD163+ macrophages, CD45+ total immune cells), and pan-CK-/CD45- stromal cells.
Number of Participants with Serious and Non-Serious Adverse Events | Baseline, 14 days to 28 days
  Grade of severity in accordance with the NCI-CTCAE version 4.0 guideline

CONTACTS AND LOCATIONS:
Overall Officials: Kimmie Ng, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No